CLINICAL TRIAL: NCT04380350
Title: Trenza Embolization Device for Intrasaccular Aneurysm Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: CDM10001446
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-02

CONDITIONS: Aneurysm; Intracranial Aneurysm
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this Post-Market Clinical Follow-up study is to assess the safety and performance of the Trenza in the treatment of intracranial aneurysms.

DETAILED DESCRIPTION:
Prospective, multi-center, single-arm, post-market follow-up study conducted in Europe for the treatment of patients with saccular intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Age is ≥18 and ≤80 years
2. Has a single, unruptured or ruptured target intracranial aneurysm that is suitable for endovascular treatment (Definition: For the purposes of this study, a ruptured intracranial aneurysm is defined as one with CT/MRI/LP evidence of subarachnoid hemorrhage attributed to the index aneurysm within the last 60 days).
3. Aneurysm morphology is saccular
4. Aneurysm size is between 6-12 mm
5. Has a wide-neck, saccular aneurysm, either bifurcation or sidewall, with a dome to neck ratio <2 or neck ≥4 mm
6. If the target intracranial aneurysm is classified as ruptured, patient must be neurologically stable with a Hunt & Hess Score of 1 or 2.
7. Must be willing to comply with protocol required procedures and follow up
8. Must be willing to sign and date an Ethics Committee approved written informed consent prior to initiation of any screening or study procedures
9. Subject or LAR must be willing to sign and date an IRB approved written informed consent prior to initiation of any screening or study procedures

Exclusion Criteria:

1. Target aneurysm has been previously treated.
2. Has significant atherosclerotic stenosis, significant vessel tortuosity, vasospasm refractory to medication, unfavorable aneurysm morphology or vessel anatomy, or some other condition(s) that, prevents or interferes with access to the target aneurysm.
3. Has undergone coiling or stenting of a non-target intracranial aneurysm within 30 days prior to study treatment or has a non-target intracranial aneurysm that is expected to be treated within 12 months following the treatment of the target aneurysm.
4. Treatment with flow diverting stent implant is anticipated.
5. A planned, staged procedure is anticipated.
6. Has Moya-Moya disease, arteriovenous malformation(s), arteriovenous fistula(e), intracranial tumor(s), intracranial hematoma(s), any other intracranial vascular malformation, or any previous major intracranial surgery.
7. Has had a recent (within 90 days) ischemic stroke, TIA, or intracranial hemorrhage.
8. Has a baseline mRS score ≥2 at time or presentation or prior to rupture (as applicable)
9. Has a known coagulopathy or is on chronic anticoagulant therapy.
10. Is pregnant or intends to become pregnant during the study or is breastfeeding.
11. Is concurrently involved in another study that could affect outcomes of IA treatment.
12. Has evidence of active cancer, terminal illness, high risk of embolic stroke, atrial fibrillation, significant co-morbidities, major surgery ≤ 30 days pre-procedure, psychiatric disorders, substance abuse, or a life expectancy of less than 5 years.
13. Has a contraindication to angiography, radiographic contrast agents, or any medications that are typically used during the procedure.
14. Patient presents a Hunt and Hess grade III or more for a ruptured aneurysm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Trenza device
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Safety primary outcome measure | 1 year (± 6 months)
  The primary safety endpoint of this study is stroke-related neurologic death, or major ipsilateral or disabling stroke in the territory supplied by the treated artery, occurring within 12 months post-procedure as adjudicated by an independent Clinical Events Committee (CEC)
  * With major ipsilateral stroke defined as a stroke associated with an increase in NIHSS score ≥ 4 points persisting ≥ 24 hours, and;
  * With disabling stroke defined as a stroke that results in a modified Rankin Scale (mRS) score ≥ 3 assessed at a minimum of 90 days post-stroke event.
Effectiveness primary outcome measure | 1 year (± 6 months)
  The primary effectiveness endpoint of this study is adequate aneurysm occlusion without retreatment or significant parent artery stenosis (>50% stenosis). The determination of adequate aneurysm occlusion using Raymond-Roy classification will be made if either of the following criteria are met:
  * 100% occlusion (Raymond Class I) demonstrated by angiographic measurement at 12 months (+6/-3 months) post-procedure, or
  * Stable Raymond Class II demonstrated on 2 serial angiographic measurements obtained a minimum of 6 months (± 1 month) apart

SECONDARY OUTCOMES:
Safety secondary outcome measure | 1 year (± 6 months)
  The secondary safety endpoint of this study is any stroke event occurring through 12 months post-procedure where a stroke event is defined as:
  • Rapidly developing clinical signs of focal (or global) disturbance of cerebral function lasting more than 24 hours with no apparent cause other than of vascular origin, including ischemic stroke and/or hemorrhagic stroke (i.e., intraparenchymal hemorrhage [IPH], subarachnoid hemorrhage [SAH], subdural hemorrhage [SDH], epidural hemorrhage [EDH]) accompanied with radiological evidence.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Cognard, Pr, Principal Investigator — Hospital Purpan, Toulouse, France
Locations (18):
- Salzburg University Hopsital, Salzburg, Austria
- Finland (2):
  - Helsinski University Hospital, Helsinki
  - Turun yliopistollinen keskussairaala, Turku
- France (6):
  - Bordeaux Hopsital, Bordeaux
  - Brest Hospital, Brest
  - HCL Lyon, Lyon
  - Montpellier Hospital, Montpellier
  - APHP Bicêtre, Paris
  - Purpan Hospital, Toulouse
- Germany (3):
  - Universitätsklinikum Knappschaftskrankenhaus Bochum GmbH, Bochum
  - Asklepios Hospital Hamburg St. Georg, Hamburg
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
- Besta hopsital, Milan, Italy
- Spain (2):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario 12 de octubre, Madrid
- United Kingdom (3):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - NHS Lothian, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow